CLINICAL TRIAL: NCT05369247
Title: Effects of Acute High-intensity Intervals Versus Moderate-intensity Continuous Cycling on Maternal and Fetal Health
Brief Title: Interval Versus Continuous Exercise During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00103630
Record Dates: First submitted 2022-03-28; First posted 2022-05-11 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2022-10

CONDITIONS: Pregnancy Related; Glucose, Low Blood; Fetal Heart Rate or Rhythm Abnormality Affecting Fetus; Fetal Blood Flow
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1st Exercise session (Experimental): Participants completed either the HIIT or MICT session.
  Interventions: Other: High intensity Interval Training; Other: Moderate Intensity Continuous Training
- 2nd Exercise session (Experimental): Participants completed the subsequent exercise protocol (i.e. HIIT or MICT)
  Interventions: Other: High intensity Interval Training; Other: Moderate Intensity Continuous Training

INTERVENTIONS:
Other: High intensity Interval Training — HIIT protocol consisted of 10 one-minute intervals of high-intensity work (i.e., > 90% HRmax) interspersed with nine one-minute intervals of self-paced active recovery (19-minutes total).
Other: Moderate Intensity Continuous Training — The MICT protocol consisted of 30-minutes of moderate intensity cycling (i.e., 64 - 76% HRmax).

SUMMARY:
The objective of this randomized cross-over design was to investigate the fetal well-being and maternal glycemic response to an acute bout of aerobic high-intensity interval training (HIIT) and moderate-intensity continuous training (MICT) with pregnant individuals.

ELIGIBILITY:
Inclusion Criteria:

* Carrying a singleton pregnancy (i.e. greater than or equal to 20 weeks of gestation).
* Has access to a stationary bike
* Located within Canada and/or within Edmonton Alberta

Exclusion Criteria:

* History of smoking within the last year
* Taking medications that may interfere with cardiovascular function.
* High-order pregnancies, e.g. twins or above.
* Females with absolute contraindications (as outlined by the Canadian Guidelines for Physical Activity throughout Pregnancy and the PARMed-X questionnaire)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Flash Glucose Monitor; interstitial Glucose | 7-days
  Measured by a Flash Glucose monitor inserted onto the back of the left tricep
Fetal Heart Rate | 3-minutes
  Measured via ultrasound pre and post exercise
Fetal Umbilical Blood Flow | 3-minutes
  Measured Via ultrasound pre and post exercise

SECONDARY OUTCOMES:
Maternal Heart Rate | 40-minutes
  Measured via heart rate monitor; Measured prior to, during, and after exercise.
Accelerometer | 7-days
  The investigators will objectively measure physical activity using an accelerometer for one week. Average number of minutes per day spent in various activity levels will be determined.
Food Log | 7-days
  The investigators will objectively measure nutrients in diet using a seven day food record. This is completed through Food Prodigy/ Food Processor software.
Perceived rating of perceived exertion | 40-minutes
  Borg Scale; Ratings from 6 - 20; Rating of six is minimal perceived exertion and rating of 20 is maximal perceived exertion.
Cardiovascular fitness | 20-minutes
  Graded exercise test to volitional fatigue.
Cerebral Blood Flow of Posterior cerebral artery | 40-min
  Measured using a trans cranial doppler ultrasound. Measured prior to, during, and after exercise.
Sleep Quality | 7-days
  The investigators will objectively measure sleep quality using an accelerometer for one week. Average number of hours of sleep per night, time spent awake after sleep onset, and number of awakenings will be determined
Rating of Perceived Enjoyment (1-10 Scale) | 40-minutes
  Rating of 1 is the lowest level of perceived enjoyment, rating of 10 is maximal perceived enjoyment
Blood pressure | 40-min
  Measured with a finometer; Measured prior to, during, and after exercise.
Cardiac Output | 40-min
  Measured with a finometer; Measured prior to, during, and after exercise.
Cerebral blood flow of middle cerebral artery | 40-minutes
  Measured using a trans cranial doppler ultrasound. Measured prior to, during, and after exercise.
fasted blood sample- sex hormones | 5-minutes
  Fasted blood samples (~30ml) will be analyzed for sex hormones (estrogen, progesterone, testosterone).
Physical Activity Questionnaire | 5-minutes
  The participants will report physical activity using the pregnancy physical activity questionnaire (gives metabolic equivalent hours per week (MET-hr/week).
Depression rating | 5-minutes
  Participants will answer a 10-question questionnaire regarding their mood. A score of 10 or higher is indicative of depressive symptoms. The investigators will report the over number of women in each group who have a score of 10+ at the start and end of the intervention.
Respiratory measures - respiratory frequency | 40-minutes
  Breathing frequency (breaths per minute). Measured using spirometry.
Respiratory measures - tidal volume | 40-minutes
  Tidal Volume (Liters per breath). Measured using spirometry.
Respiratory measures - oxygen | 40-minutes
  Oxygen metabolism (% oxygen used per breath). Measured using a gas analyzer.
Respiratory measures - carbon dioxide | 40-minutes
  Carbon Dioxide production (% carbon dioxide per breath). Measured using a gas analyzer.
Respiratory measures - lung volume | 40-minutes
  Total Lung Capacity (Liters). Measured using spirometry.
Fetal Outcome - birth weight | within one month postpartum
  Participants will provide the investigators with birth weight for the infant (grams)
fetal outcomes- length | within one month postpartum
  Participants will provide the investigators with birth length for the infant (cm)
fetal outcomes- gestational age | within one month postpartum
  Participants will provide the investigators with gestational age at delivery (weeks)
maternal outcomes- mode of delivery | within one month postpartum
  Participants will provide the investigators with mode of delivery (vaginal or cesarean).
maternal outcomes- delivery complications | within one month postpartum
  Participants will provide the investigators with information regarding any delivery complications.
maternal outcomes- pregnancy complications | any time during study
  Participants will provide the investigators with information regarding any pregnancy complications (gestational diabetes, pregnancy induced hypertension, preeclampsia).
fetal outcomes- NICU | within one month postpartum
  Participants will provide the investigators with information regarding length (days) of admission to Neonatal Intensive Care Unit (NICU) if applicable
maternal outcomes- gestational weight gain | within one month postpartum
  Participants will provide the investigators with the last maternal weight immediately before delivery. This will be used to calculate gestational weight gain (kg; last maternal weight - self reported pre-pregnancy weight).

CONTACTS AND LOCATIONS:
Overall Officials: Margie H Davenport, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Wowdzia JB, Hazell TJ, Berg ERV, Labrecque L, Brassard P, Davenport MH. Maternal and Fetal Cardiovascular Responses to Acute High-Intensity Interval and Moderate-Intensity Continuous Training Exercise During Pregnancy: A Randomized Crossover Trial. Sports Med. 2023 Sep;53(9):1819-1833. doi: 10.1007/s40279-023-01858-5. Epub 2023 May 22. PMID 37213048